CLINICAL TRIAL: NCT05285072
Title: Siderophores for Imaging Infection: A First-in-human Pilot Study Using a Tracer (68Ga-DFO) as Proof of Concept That Siderophores Can Image Bacterial Infection in Vascular Grafts
Brief Title: Siderophores for Imaging Infection Using 68Ga-DFO
Acronym: GaDFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 271229
Record Dates: First submitted 2021-02-02; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Vascular Graft Infection
Keywords: positron emission tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vascular graft infection: Patients with confirmed vascular graft infection according to current syndromic criteria.
  Interventions: Radiation: PET-CT scan
- Vascular graft without infection: Patients with no clinical evidence of infection and CRP less than 5.
  Interventions: Radiation: PET-CT scan

INTERVENTIONS:
Radiation: PET-CT scan — PET-CT scan using 68Ga-DFO

SUMMARY:
This is a single center pilot study involving a single study visit for participants, with remote follow up data collected at 24 hours. Follow up at 3 months and 6 months later occurs as standard of care.

The purpose of the study is to find out if a new type of imaging tracer (68Ga-DFO) can be used to show infection in patients with vascular grafts using PET/CT scans. These infections may be associated with significant ill health and mortality and can be difficult to diagnose. Effective treatments can require major surgery and long-term antibiotic therapy which may not be well tolerated nor feasible. Development of new imaging tracers that could detect bacteria causing graft infections with PET-CT scanners has great potential to benefit patients being considered for vascular surgery.

A PET-CT scan combines images from a CT (Computerised Tomography) scan and a PET (Positron Emission Tomography) scan. The CT scan takes a series of X-rays across the organs inside the body. The PET scan uses a mildly radioactive tracer to show up areas of activity inside the body. The 68Ga-DFO tracer mimics particles that bacteria make to take up iron from the body to help them grow. The investigators hope this new tracer will go to areas where bacteria are causing infection and tell if the graft is infected. The investigators hope this type of tracer could be a better way to show infection than the tests currently used to diagnose infection.

DETAILED DESCRIPTION:
This study is a first in human mechanistic study hypothesizing that siderophore complexes labelled with a radiotracer (Gallium-68) will be taken up in sites of infection in patients with a vascular graft.

Study objectives are to:

i) Determine if siderophore uptake occurs in sites of infection using the radiolabelled siderophore 68Ga-DFO in patients with a vascular graft on PET/CT scans.

ii) Determine if siderophore uptake as measured by the radiolabelled siderophore 68Ga-DFO is specific for infection by exploring whether uptake occurs in individuals with vascular grafts without infection and by characterising the uptake in normal tissues.

The injected substances are well-known licensed products.

The study will involve performing 68Ga-DFO PET/CT scans in 30 patients with vascular grafts, including 25 patients with diagnosed infection according to current syndromic criteria and 5 patients with a vascular graft but no evidence of any infection. Patients with infection will be recruited from patients who have had a prior FDG-PET-CT scan performed as part of their routine care which shows suspected graft infection.

All patients will have 'static' PET-CT scans following injection of the tracer. The scans will take 30 minutes.

The first ten patients with graft infection will also have 'dynamic' scans performed immediately after tracer injection lasting for 90 minutes. The result of these scans (e.g. time activity curves) will inform the scan protocol of the subsequent patients (e.g. uptake time). Up to 10 of these patients will have venous blood sampling at 8 time points up to 120 minutes after injection.

Patients will be followed up in person or by telephone 24 hours after the scan. Apart from this no specific follow up procedure outside standard of care is planned within this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Women of childbearing potential must have documented negative pregnancy test prior to tracer administration.
* Willing and able to give informed consent
* Able to comply with the PET imaging protocol
* Patients with vascular grafts in situ
* Positive FDG-PET/CT in the case of patients with suspected or diagnosed graft infections

Exclusion Criteria:

* Aged under 18
* Pregnancy or lactation
* Prisoners
* Any lack of capacity to consent, including lack of adequate understanding of written or spoken English.
* Iron infusion within 1 week of 68Ga-DFO PET/CT scan (can potentially hamper the sensitivity of DFO by decreasing the number of siderophore receptors in the bacteria).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cohort 1 Patients attending the Department of Vascular Surgery or the PET Centre (after referral for a PET scan with the indication of suspected or diagnosed vascular graft infection) at Guy's & St. Thomas' Hospitals in London.
  Cohort 2 Patients with no evidence of vascular graft infection attending a routine follow-up visit after surgery in the Department of Vascular Surgery at Guy's & St. Thomas' Hospitals . Patients will have a blood sample prior to imaging to ensure that CRP is ≤5.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
siderophore uptake | baseline
  Observe level of siderophore uptake around vascular graft in patients with known infection and in patients without infection

SECONDARY OUTCOMES:
Infective agents associated with a confirmed vascular graft infection | 6 months post baseline
  from blood cultures or organisms recovered from an explanted graft, intra-operative specimen, from percutaneous or radiologically guided aspirate of peri-graft fluid

OTHER OUTCOMES:
Infection diagnosis | 6 months post baseline
  Details will be collected of any evidence of vascular graft infection from blood cultures or organisms recovered from an explanted graft, intra-operative specimen, from percutaneous or radiologically guided aspirate of peri-graft fluid and therapy received.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Barrington, MD, Principal Investigator — King's College London
Locations (1):
- Kings College London and Guy's and St Thomas' Hospital PET Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No